CLINICAL TRIAL: NCT05347563
Title: Study on Ventilation Distribution With Electrical Impedance Tomography for Paediatric Respiratory Failure: Impact of Intervention
Brief Title: Study on Ventilation Distribution With Electrical Impedance Tomography for Paediatric Respiratory Failure
Acronym: PELUCHE1
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0111; 2022-A00505-38 (Other: IDRCB)
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure
Keywords: Electrical impedance tomography; Children; Pediatric intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: group A: Patient < 18 years old admitted to a continuous monitoring unit - resuscitation for acute respiratory failure regardless of the ventilation modality and benefiting from TIE monitoring
  Interventions: Procedure: Electrical impedance tomography
- Group B (reference): Group B (reference): Patient under general anesthesia with mechanical ventilation without respiratory pathology.
  Interventions: Procedure: Electrical impedance tomography

INTERVENTIONS:
Procedure: Electrical impedance tomography — All change in ventilator settings (mode, tidal volume or inspiratory pressure, Peep, recruitment…)

SUMMARY:
Electrical impedance tomography (EIT) is a non-invasive, bedside monitoring technique that provides continuous, real-time information about the regional distribution of the ventilation.

There are very few data in children admitted to the PICU (pediatric intensive care unit) and the aim of the study is to describe the distribution of the ventilation in children with acute respiratory failure and to study the impact of the interventions in the PICU (change in ventilatory settings, change in position, suction, respiratory kinesiotherapy,…)

DETAILED DESCRIPTION:
Children with acute respiratory failure admitted to the PICU (pediatric intensive care unit)

ELIGIBILITY:
Inclusion Criteria:

Groupe A

* children < 18 years
* Admitted to the PICU with acute respiratory failure
* Monitoring with EIT
* non opposition of parents or legal representative Groupe B
* children < 18 years
* With general anesthesia and mechanical ventilation
* Monitoring with EIT
* non opposition of parents or legal representative

Exclusion Criteria:

* Monitor not available
* contra indication to the use of thoracic belt
* Intraoperative period with use of electrocautery
* Child not affiliated to a social security system and under protective measures legal

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 250 Childrens group A: Patient < 18 years old admitted to a continuous monitoring unit - resuscitation for acute respiratory failure regardless of the ventilation modality and benefiting from TIE monitoring Group B (reference): Patient under general anesthesia with mechanical ventilation without respiratory pathology.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Distribution of Ventilation | up to 48 hours
  Distribution of ventilation as determined by changes in impedence in region of interest

CONTACTS AND LOCATIONS:
Overall Officials: Florent Baudin, MD, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Hôpital Femme Mère Enfant Service de néonatologie et réanimation néonatale, Bron, Rhone
  - Hôpital Femme Mère Enfant Service de réanimation et d'urgence pédiatrique, Bron, Rhone
  - Paediatric intensive care Unit, Bron, Rhone
  - Hôpital Louis Pradel GHE - Réanimation Cardiaque Pédiatrique (U11), Bron, Rhone

IPD SHARING:
Plan to Share IPD: No